CLINICAL TRIAL: NCT04047368
Title: Comparison of Coronary Lithoplasty and Rotablation for the Interventional Treatment of Severely Calcified Coronary Stenoses - ROTA.Shock-Trial
Brief Title: Comparison of Coronary Lithoplasty and Rotablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Else Kröner-Fresenius Stiftung, Bad Homburg, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROTA.shock
Record Dates: First submitted 2019-07-22; First posted 2019-08-06 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Calcified Atheroma
Keywords: Percutaneous coronary intervention; Rotablation; Coronary lithoplasty; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotablation (Active Comparator)
  Interventions: Procedure: Rotablation
- Coronary Lithoplasty (Experimental)
  Interventions: Procedure: Coronary Lithoplasty

INTERVENTIONS:
Procedure: Rotablation — Percutaneous Coronary Intervention using Rotablation
  Arms: Rotablation
Procedure: Coronary Lithoplasty — Percutaneous Coronary Intervention using Lithoplasty
  Arms: Coronary Lithoplasty

SUMMARY:
This study compares a new method of treating severely calcified coronary lesions, the intracoronary lithoplasty, with the current gold standard, the rotablation.

DETAILED DESCRIPTION:
Severe coronary calcification is still a challenge for percutaneous coronary intervention (PCI). Reduction of the calcified plaque mass is necessary to achieve adequate stent expansion during further course. Rotablation has been the only reliable option to treat extremely calcified coronary lesions for a long time. Coronary lithoplasty has been recently introduced as a new promising treatment option in this special subset. It provides the unique opportunity to break severely calcified plaque structures even inside deeper layers of the vessel wall. Aim of this study is to compare rotablation and coronary lithotripsy for treatment of severely calcified coronary lesions. Plaque structure, plaque volume, as well as lumen diameters will be analyzed by optical coherence tomography (OCT) before and after debulking, as well as after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 yrs
* Stable coronary heart disease or acute coronary syndromes
* Single or multi vessel disease. Vessel is defined as, left anterior descending, left circumflex, and right coronary arteries. Any branch within the vessel is considered part of the vessel.
* Written informed consent was obtained before the procedure
* Severely calcified coronary lesion with indication for rotablation

Exclusion Criteria:

* Known renal insufficiency (serum creatinine clearance <30ml/min/1.73m² or receiving dialysis)
* Known allergy against protocol-required medications including ASS, prasugrel, ticagrelor, clopidogrel, heparin. History of bleeding diathesis or known coagulopathy
* Cardiogenic shock
* Lesion length > 32mm
* Bifurcation lesions requiring 2-Stent-Strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Minimal Stent Area (End of the Procedure) | 0 days

SECONDARY OUTCOMES:
Minimal/Mean/Maximal Stent Diameter | 0 days
Minimal/Mean/Maximal Lumen area | 0 days
Minimal/Mean/Maximal Lumen diameter | 0 days
Mean/Maximal Stent area | 0 days
Incidence of target lesion failure | 0 months; 1 month; 6 months
Incidence of target vessel failure | 0 months; 1 month; 6 months
MACE rate | 0 months; 1 month; 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Florian Blachutzik, Dr., Principal Investigator — University of Giessen
Locations (1):
- University of Giessen, Giessen, Germany

REFERENCES:
- [Derived] Blachutzik F, Meier S, Weissner M, Schlattner S, Gori T, Ullrich-Daub H, Gaede L, Achenbach S, Mollmann H, Chitic B, Aksoy A, Nickenig G, Weferling M, Dorr O, Boeder N, Bayer M, Elsasser A, Hamm C, Nef H; ROTA.Shock Investigators. Comparison of Coronary Intravascular Lithotripsy and Rotational Atherectomy in the Modification of Severely Calcified Stenoses. Am J Cardiol. 2023 Jun 15;197:93-100. doi: 10.1016/j.amjcard.2023.02.028. Epub 2023 Apr 2. PMID 37012181